CLINICAL TRIAL: NCT03289559
Title: Testosterone Effects on Systemic Lipolysis and Whole Body Lipid Utilization
Brief Title: Effects of Testosterone and Fat Utilization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 06-0010
Record Dates: First submitted 2017-09-18; First posted 2017-09-21 (Actual); Last update posted 2017-09-21 (Actual); Status verified 2017-09

CONDITIONS: Healthy; Volunteers
MeSH Terms: interventions — LHRH, Ac-Nal(1)-Cpa(2)-Trp(3)-Arg(6)-Ala(10)-; Aromatase Inhibitors

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention)
- GnRH antagonist + Placebo Gel (Placebo Comparator)
  Interventions: Drug: GnRH antagonist; Drug: Aromatase Inhibitors
- GnRH antagonist + Testosterone Gel (Active Comparator)
  Interventions: Drug: GnRH antagonist; Drug: Aromatase Inhibitors; Drug: Testosterone gel

INTERVENTIONS:
Drug: GnRH antagonist
  Arms: GnRH antagonist + Placebo Gel; GnRH antagonist + Testosterone Gel
Drug: Aromatase Inhibitors
  Arms: GnRH antagonist + Placebo Gel; GnRH antagonist + Testosterone Gel
Drug: Testosterone gel
  Arms: GnRH antagonist + Testosterone Gel

SUMMARY:
Evidence is accumulating that there are sex differences in energy and substrate metabolism. The positive or negative consequences of such metabolic differences between men and women need to be evaluated with respect to health outcomes. The importance of aberrant lipid metabolism in metabolic diseases such as obesity, diabetes and cardiovascular disease, makes understanding the distinction between "normal" vs aberrant critical to future treatment and prevention strategies. Sex differences in the effects of catecholamines on lipid metabolism and substrate oxidation in non-obese, healthy individuals, have been consistently observed. In addition, distinct differences in men and women exist in the distribution of body fat, with men typically having greater central adiposity than women. Accumulation of fat in the abdomen is associated with an increased risk for metabolic abnormalities such as hyperlipidemia and insulin resistance. In the current study, therefore, the role of testosterone in determining the sex differences in catecholamine mediated substrate metabolism and deposition of dietary fat into upper versus lower body adipose tissue depots will be addressed.

ELIGIBILITY:
Inclusion Criteria:

* normal weight (BMI of 23-29.9 kg/m2)
* not be highly trained (< 5hrs of moderate intensity, planned exercise per week).

Exclusion Criteria:

* Patients will be excluded if they have one or more of the following out-of-range values measured on a fasting blood sample:
* glucose <65 or > 110 mg/dl,
* insulin > 20 uU/ml,
* thyroid stimulating hormone <0.5 or >5.0 uU/ml,
* growth hormone >2.5 ng/ml.
* Subjects who may be:
* anemic (hemoglobin < 14.5 g/dl men ),
* have abnormal liver function tests:

  * alanine amino transferase > 47 U/l,
  * aspartate aminotransferase, > 47 U/l,
  * alkaline phosphatase <39 or >117 U/l) or
  * creatinine (<0.6 or >1.1 mg/dl).

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2006-01-01 (Actual); Primary Completion 2011-01-01 (Actual); Study Completion 2014-01-01 (Actual)

PRIMARY OUTCOMES:
Dietary fat tracer for storage of meal derived fatty acids | 4 weeks
  50 uCi of [1-14C] oleic acid administered with an inpatient test meal

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Bessesen, MD, Principal Investigator — University of Colorado, Denver

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rynders CA, Schmidt SL, Bergouignan A, Horton TJ, Bessesen DH. Effects of short-term sex steroid suppression on dietary fat storage patterns in healthy males. Physiol Rep. 2018 Jan;6(2):e13533. doi: 10.14814/phy2.13533. PMID 29380951